CLINICAL TRIAL: NCT01095081
Title: GARDIAN, Gadovist in Routine Diagnostic Magnetic Resonance Imaging Administration in Non-selected Patients
Acronym: GARDIAN
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14823; GV0901 (Other: company internal)
Record Dates: First submitted 2010-03-17; First posted 2010-03-29 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Magnetic Resonance Imaging; Magnetic Resonance Angiography
MeSH Terms: interventions — gadobutrol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Gadobutrol (Gadovist, BAY86-4875)

INTERVENTIONS:
Drug: Gadobutrol (Gadovist, BAY86-4875) — Patients requiring contrast enhanced MRI using Gadovist. Administration of Gadovist at the discretion of the attending physician.

SUMMARY:
Prospective, non-interventional, multi-center study. The observation period for each subject covers the treatment period with Gadovist®. For each patient, the treating physician or nurse documents demographics, medical data, safety parameters and treatment signs and symptoms at the visit. Patients with severe renal impairment will be followed-up after 3 month by phone call from the investigator if in line with routine practice. Data audit/monitoring by source data verification will be done in a subset of sites and patients

DETAILED DESCRIPTION:
Evaluate the safety and tolerability of Gadovist in patients requiring contrast-enhanced MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing contrast enhanced Magnetic Resonance Imaging with Gadobutrol (Gadovist).

Exclusion Criteria:

* There are no other exclusion criteria beyond the contraindications contained in the Summary of Product Characteristics (hypersensitivity to the active substance or to any of the excipients) and the warnings.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Evaluate the safety and tolerability of Gadovist in patients requiring contrast-enhanced MRI.
Sampling Method: Non-Probability Sample
Enrollment: 23775 (Actual)
Dates: Start 2010-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Event Collection / Calculation of Adverse Event rates in Study population and subgroups | 1 day

SECONDARY OUTCOMES:
Analysis of Adverse Event Collection rates according to age, gender, concomitant diseases and risk factors, dose administered. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (20):
- Many Locations, Bosnia and Herzegovina
- Many Locations, Canada
- Many Locations, China
- Many Locations, Czechia
- Many Locations, France
- Many Locations, Germany
- Many Locations, Greece
- Many Locations, Hong Kong
- Many Locations, Hungary
- Many Locations, Italy
- Many Locations, Kazakhstan
- Many Locations, Kyrgyzstan
- Many Locations, Poland
- Many Locations, Russia
- Many Locations, South Africa
- Many Locations, South Korea
- Many Locations, Spain
- Many Locations, Taiwan
- Many Locations, Thailand
- Many Locations, Vietnam